CLINICAL TRIAL: NCT03154294
Title: A Phase 1 Evaluation of the Safety and Tolerability of TAK-228 in Combination With TAK-117 and Paclitaxel in Advanced Solid Tumors
Brief Title: Evaluation of the Safety and Tolerability of TAK-228 With TAK-117 and Paclitaxel in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: X31025
Record Dates: First submitted 2017-05-08; First posted 2017-05-16 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-02

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Paclitaxel; sapanisertib; serabelisib

STUDY DESIGN:
Intervention Model Description: The demographic and clinical characteristics of the study patients will be summarized using descriptive statistics
  * Primary objective: The maximum tolerable dose will be assessed, which is the dose level at which < one-third of patients will experience a dose-limiting toxicity
  * Secondary objectives:
    1. Adverse events will be defined according to the Common Terminology Criteria for Adverse Events v4 and will be summarized with descriptive statistics
    2. Response rate will be determined according to the Response Evaluation Criteria in Solid Tumors 1.1 response criteria. Number and type of responses will be summarized with descriptive statistics
  * Exploratory objectives
    1. Response rate and relationship with genomic alterations will be examined by using a two-sided Fisher Exact test due to the small sample sizes
    2. Therapy-Related Symptom Checklist and Health-Related Quality of Life Linear Analogue Self-Assessment scores will be summarized with descriptive statistics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Paclitaxel 60mg/m2 Day 1, Day 8, Day 15 TAK-228 2mg Days 2-4, Days 9-11, Days 16-18, Days 23-25 TAK-117 100mg Days 2-4, Days 9-11, Days 16-18, Days 23-25
  Interventions: Drug: paclitaxel; Drug: TAK-228; Drug: TAK-117
- Cohort 2 (Experimental): Paclitaxel 60mg/m2 Day 1, Day 8, Day 15 TAK-228 2mg Days 2-4, Days 9-11, Days 16-18, Days 23-25 TAK-117 200mg Days 2-4, Days 9-11, Days 16-18, Days 23-25
  Interventions: Drug: paclitaxel; Drug: TAK-228; Drug: TAK-117
- Cohort 3 (Experimental): Paclitaxel 80mg/m2 Day 1, Day 8, Day 15 TAK-228 2mg Days 2-4, Days 9-11, Days 16-18, Days 23-25 TAK-117 200mg Days 2-4, Days 9-11, Days 16-18, Days 23-25
  Interventions: Drug: paclitaxel; Drug: TAK-228; Drug: TAK-117
- Cohort 4 (Experimental): Paclitaxel 80mg/m Day 1, Day 8, Day 15 TAK-228 3mg Days 2-4, Days 9-11, Days 16-18, Days 23-25 TAK-117 200mg Days 2-4, Days 9-11, Days 16-18, Days 23-25
  Interventions: Drug: paclitaxel; Drug: TAK-228; Drug: TAK-117
- Cohort 5 (Experimental): Paclitaxel 80mg/m2 Day 1, Day 8, Day 15 TAK-228 4mg Days 2-4, Days 9-11, Days 16-18, Days 23-25 TAK-117 200mg Days 2-4, Days 9-11, Days 16-18, Days 23-25
  Interventions: Drug: paclitaxel; Drug: TAK-228; Drug: TAK-117

INTERVENTIONS:
Drug: paclitaxel — Paclitaxel will be diluted prior to infusion in 0.9% Sodium Chloride for Injection, USP; 5% Dextrose Injection, USP; 5% Dextrose and 0.9% Sodium Chloride Injection, USP; or 5% Dextrose in Ringer's Injection to a final concentration of 0.3 to 1.2mg/mL. At ambient temperature (approximately 25°C) and room lighting conditions the solution is physically and chemically stable for up to 27 hours. The diluted product will be prepared and stored in glass, polypropylene, or polyolefin containers; DEHP-containing (polyvinyl chloride (PCV)) containers should not be used. Paclitaxel will be administered using a vented Paclitaxel set with in-line 0.22-micron filter and run over 1 hour.
  Other Names: Taxol
Drug: TAK-228 — TAK-228 will be provided in 30-ct, 60-cc high density polyethylene (HDPE) bottles with polypropylene, child-resistant caps and induction seal. TAK-228 will be administered on an empty stomach. It is recommended that each dose of TAK-228 + TAK-117 be given PO with 8 ounces (240 mL) of water. Patients should be instructed to refrain from eating and drinking (except for water and prescribed medications) for 2 hours before and 1 hour after each dose.
  Other Names: INK128; MLN0128
Drug: TAK-117 — TAK-117 will be provided in 30-ct, 60-cc high density polyethylene (HDPE) bottles with polypropylene, child-resistant caps and induction seal. TAK-117 will be administered on an empty stomach. It is recommended that each dose of TAK-228 + TAK-117 be given PO with 8 ounces (240 mL) of water. Patients should be instructed to refrain from eating and drinking (except for water and prescribed medications) for 2 hours before and 1 hour after each dose.
  Other Names: MLN1117; INK1117

SUMMARY:
This is an open-label, cohort study to determine the feasibility and tolerability of the combination of TAK-228 and TAK-117 given on days 2-4, 9-11, 16-18, and 23-25 with paclitaxel on days 1, 8, and 15 for one 28-day cycle in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The goal of this study is to determine a tolerated dose of the combination of TAK-228, TAK-117 and paclitaxel. To do this, investigators will estimate the maximum tolerated dose that is defined as the dose level at which less than one-third of patients will experience a dose-limiting toxicity. A traditional dose escalation design will be used, beginning with the lowest dose level and escalating to the maximum allowable dose level as specified in the protocol. Three patients will be treated one at a time at a given dose level. A maximum of 5 dosing levels results in a maximum sample size of n=30 subjects. Adverse events will be defined using the Common Toxicity Criteria v. 4.0. dose-limiting toxicity is defined as:

* Grade 3 or higher nonhematologic toxicity, despite adequate treatment, except for the following:

  * Grade 3 hyperglycemia lasting ≤14 days (all patients should receive optimal antiglycemic treatment, including insulin, as clinically indicated).
  * Grade 3 rash lasting ≤3 days (all patients should receive topical steroid treatment, oral antihistamines, and oral steroids, if necessary).
  * Inadequately treated Grade 3 nausea and/or vomiting and Grade 3 diarrhea (all patients should receive optimal antiemetic and/or antidiarrheal prophylaxis and/or treatment).
* Grade 4 neutropenia lasting >7 days in the absence of growth factor support.
* Grade 4 neutropenia of any duration accompanied by fever ≥38.5°C and/or systemic infection.
* Any other ≥Grade 4 hematologic toxicity.
* Inability to administer at least 75% of planned doses of TAK-228 within Cycle 1, due to study drug-related toxicity.
* Any clinically significant occurrence that the investigator and sponsor agree would place patients at an undue safety risk.

Patients experiencing any grade 3 or more hematologic toxicity attributed to the treatment will hold all therapy until resolution of the toxicity to grade 2 or less. If toxicity persists, the patients will be removed from the study. Upon resolution of the toxicity, the patient will restart treatment at the original dose at the discretion of the investigators.

One of the following outcomes will determine the treatment of subsequent patients:

* If none of the three patients experiences a dose-limiting toxicity, the next group of patients will be entered in the next higher dose cohort. All patients within a cohort must have completed at least once cycle (28 days) prior to initiation of the next cohort of patients.
* If one of the three patients experiences a dose-limiting toxicity, three more patients will be accrued at the current dose level. Subsequently, if only one of the six patients treated at this level experiences a dose-limiting toxicity, the dose will be escalated to the next higher dose in the next group of patients. If two or more of the six patients experiences a dose-limiting toxicity, the maximum tolerated dose has been exceeded and is defined as the previous dose at which no more than 1/3 experienced a dose-limiting toxicity.
* If at least two of the three experience a dose-limiting toxicity, the maximum tolerated dose has been exceeded and is defined as the previous dose at which no more than 1/3 experienced a dose-limiting toxicity.

If the lowest allowable dose level exceeds the maximum tolerated dose, the study will be terminated and the combination will not be deemed safe for use in this population. Additionally, the highest dose level will not be exceeded, even if no dose-limiting toxicities are experienced at that dose.

The adverse events overall and by individual adverse events categories will be summarized. Serious adverse events will be summarized in a similar manner. These summaries will be performed overall and for each dose cohort. Investigators will summarize all events as well as the highest grade for a given subject. Investigators will summarize the number of subjects that exhibit a dose-limiting toxicity at each dose cohort and describe the dose-limiting toxicity for each subject, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older
* Patients must have a diagnosis of an advanced solid tumor malignancy and must be refractory to or intolerant of existing therapies known to provide a clinical benefit
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status of 0-2
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential must have a negative pregnancy test and agree to practice one effective method of pregnancy prevention contraception and one additional effective (barrier) method, at the same time, from the time of signing the informed consent through 90 days (or longer as mandated by local labeling [e.g., USPI, SmPC, etc.,]) after the last dose of study drug, OR
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, sympto- thermal and post ovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:

  * Agree to practice highly effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, OR
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, sympto- thermal and post ovulation methods for the female partner], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
  * Agree not to donate sperm during the course of this study or within 120 days after receiving their last dose of study drug
* Screening clinical laboratory values as specified below:

  * Bone marrow reserve consistent with: absolute neutrophil count (ANC) ≥1.5 x 109/L; platelet count ≥100 x 109/L; hemoglobin ≥9 g/dL without transfusion within 1-week preceding study drug administration
  * Hepatic: total bilirubin ≤1.5 x upper limit of normal (ULN), transaminases (aspartate aminotransferase/serum glutamic oxaloacetic transaminase- AST/SGOT and alanine aminotransferase/serum glutamic pyruvic transaminase-ALT/SGPT) ≤2.5 x ULN (≤5 x ULN if liver metastases are present)
  * Renal: creatinine clearance ≥50 mL/min based either on Cockcroft-Gault estimate or based on urine collection (12 or 24 hour)
  * Metabolic: Glycosylated hemoglobin (HbA1c) <7.0%, fasting serum glucose (≤ 130 mg/dL) and fasting triglycerides ≤300 mg/dL
* Ability to swallow oral medications
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that the patient may withdraw consent at any time without prejudice to future medical care
* Patients who have a history of brain metastasis are eligible for the study provided that all the following criteria are met:

  * Brain metastases which have been treated
  * No evidence of disease progression for ≥3 months before the first dose of study drug
  * No hemorrhage after treatment
  * Off-treatment with dexamethasone for 4 weeks before administration of the first dose of TAK-228
  * No ongoing requirement for dexamethasone or anti-epileptic drugs

Exclusion Criteria:

* Active central nervous system (CNS) metastasis
* Other clinically significant co-morbidities, in the opinion of the investigators, such as uncontrolled pulmonary disease, active central nervous system disease, active infection, or any other condition that could compromise the patient's participation in the study
* Known human immunodeficiency virus infection
* Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Diagnosed or treated for another malignancy within 2 years before administration of the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Breast feeding or pregnant
* Treatment with any investigational products within 30 days before the first dose of study drug
* Previous treatment with PI3K, AKT, dual PI3K/mTOR inhibitors, TORC1/2 inhibitors (prior treatment with everolimus is allowed)
* Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of TAK-228. In addition, patients with small bowel or jejunal stomata are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2022-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Casey Williams, PharmD, Principal Investigator — Avera Cancer Institute
Locations (1):
- Avera Cancer Institute, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Starks DC, Rojas-Espaillat L, Meissner T, Williams CB. Phase I dose escalation study of dual PI3K/mTOR inhibition by Sapanisertib and Serabelisib in combination with paclitaxel in patients with advanced solid tumors. Gynecol Oncol. 2022 Sep;166(3):403-409. doi: 10.1016/j.ygyno.2022.07.005. Epub 2022 Jul 15. PMID 35843739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at Avera Cancer Institute in Sioux Falls, South Dakota, United States from July 2017 to April 2020.
Pre-assignment Details: A total of 19 participants with a diagnosis of an advanced solid tumor malignancies were enrolled in this study.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 4 | 3 | 3 | 6 | 3
Completed | 4 | 3 | 3 | 4 | 2
Not Completed | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 3 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 4 | 1 | 11
  >=65 years | 2 | 1 | 1 | 2 | 2 | 8
Age, Continuous [Median (Full Range); unit: years] | 65.25 [59.3 to 75.4] | 63.9 [56.1 to 66.6] | 61.8 [61.4 to 69.6] | 64.55 [56.3 to 68.2] | 66.6 [48.9 to 72.4] | 64.7 [48.9 to 75.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 6 | 3 | 19
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 6 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Developed Does-limiting Toxicity (DLT)
Description: DLT is defined as any death not clearly due to underlying disease or extraneous causes; critical liver injury by Hy's Law; grade 3 or higher toxicity (with certain exceptions); inability to administer at least 75% of planned doses of TAK-228 within Cycle 1, due to study drug-related toxicity and any other clinically significant occurrence that the investigator and sponsor agree would place patients at an undue safety risk.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 5: Paclitaxel 80mg/m2 Day 1, Day 8, Day 15TAK -228 4mg Days 2-4, Days 9-11, Days 16-18, Days 23-25 TAK-117 200mg Days 2-4, Days 9-11, Days 16-18, Days 23-25
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 3
Participants | 0 | 0 | 0 | 0 | 1

2. Secondary Outcome: Number of Patients With Beneficial Clinical Response
Description: Tumor objective response is assessed by CT or MRI and evaluated according to RECIST 1.1 response criteria. Complete Response (CR, disappearance of all target lesions), partial response (PR, >= 30% decrease of target lesions) and stable disease (SD, either the increase of target lesion is less than 20% or not sufficient shrinkage to qualify for PR) are considered as beneficial clinical response.
Time Frame: 27 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 4 | 1 | 3 | 4 | 3
Participants | 3 | 1 | 2 | 3 | 2

3. Secondary Outcome: Number of Patients With Tumor Objective Response
Description: Tumor objective response is assessed by CT or MRI and evaluated according to RECIST 1.1 response criteria. Complete Response (CR, disappearance of all target lesions) and partial response (PR, >= 30% decrease of target lesions) are considered as beneficial clinical responses.
Time Frame: 27 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 4 | 1 | 3 | 4 | 3
Participants | 2 | 1 | 1 | 2 | 1

4. Secondary Outcome: Progression Free Survival (in Month)
Description: Tumor assessment according to RECIST 1.1 was performed at the end of the third cycle, and then every 12 week until study discontinuation or disease progression, whichever is later. For those patients without disease progression at the end of therapy, tumor assessments were undertaken every 3 month until either disease progression os observed or further anti-cancer treatment is initiated.
Time Frame: 27 months
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 1 | 2 | 3 | 2
months | 10 [9 to 11] | 19 [19 to 19] | 6 [6 to 6] | 10 [4 to 13] | 17 [7 to 27]

5. Secondary Outcome: Overall Survival
Description: All patients were contacted for survival status following study discontinuation at 4, 8, 12,18 and 24 months.
Time Frame: Baseline until date of death, assessed up to 43 months
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 3
months | 18 [12 to 20] | 9 [5 to 43] | 13 [5 to 26] | 8 [3 to 29] | 23 [12 to 27]

6. Other Pre Specified Outcome: Number of Patients With MTOR and PI3K Alterations Who Had Clinical Favorable Responses.
Description: as for outcome 2
Time Frame: 27 months
Population: Only patients with genomic alteration at MTOR and PIK3CA are analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 2 | 0 | 2 | 1
Participants | 1 | 1 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and Other (Not Including Serious) Adverse Events were collected up to 27 months. All-Cause Mortality was collected up to 43 months.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 4/4 | 2/3 | 3/3 | 6/6 | 2/3
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/3 | 1/3 | 6/6 | 3/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=6) | Cohort 5 (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 2 (9) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
General disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Worsened Ventral Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (2) | 1 (2) | 3 (4) | 2 (4)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
White blood cell decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 2 (5) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 1 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=6) | Cohort 5 (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (7) | 1 (5) | 1 (4) | 6 (23) | 3 (16)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 2 (3) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Fatigue (General disorders) | 2 (4) | 1 (3) | 2 (5) | 5 (8) | 3 (6)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2) | 5 (15) | 3 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Worsened Ventral Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (5) | 0 (0) | 1 (3) | 5 (11) | 3 (6)
Nausea (Gastrointestinal disorders) | 4 (7) | 2 (4) | 3 (4) | 5 (8) | 3 (10)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (3) | 1 (2) | 0 (0) | 4 (6) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (7) | 0 (0) | 1 (1) | 3 (4) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (4) | 3 (8) | 1 (3) | 3 (3) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (2) | 1 (1) | 1 (2) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (5) | 1 (1) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (2)
Neutrophil count decreased (Investigations) | 3 (4) | 2 (10) | 2 (7) | 5 (23) | 3 (12)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 2 (7)
Weight loss (Investigations) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 2 (2)
White blood cell decreased (Investigations) | 4 (18) | 3 (15) | 3 (8) | 5 (32) | 3 (33)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (5) | 2 (3) | 2 (5) | 5 (10) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (7) | 0 (0) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3) | 1 (1) | 3 (9) | 3 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (8) | 1 (2) | 1 (1) | 4 (12) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (15) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 2 (10)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain (Tailbone) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (2) | 2 (2)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 3 (4) | 0 (0) | 0 (0) | 4 (5) | 2 (3)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (2) | 3 (5) | 2 (5)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (2) | 3 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bloody Sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 2 (3) | 5 (9) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT03154294/Prot_SAP_000.pdf